CLINICAL TRIAL: NCT04006886
Title: Gluten-free Diet in Patients With Primary Sclerosing Cholangitis (PSC) - a Pilot-Study
Brief Title: Gluten-free Diet in Patients With Primary Sclerosing Cholangitis (PSC)
Acronym: PSt-GFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Institute for Clinical Molecular Biology, Christian-Albrechts-University, Kiel (Unknown); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marcus Tetzlaff, study coordinator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSt-GFD
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Reduction of Intestinal Inflammatory Activity
MeSH Terms: interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — After run-in phase with normal diet under Observation, patients will be on a gluten-free diet for two months.

SUMMARY:
Gluten is a protein found in wheat and other cereals as barley and rye. It triggers an inflammatory reaction in the small-bowel of genetically predisposed persons. Alpha-amylase/trypsin inhibitors (ATIs) of wheat seem to be the responsible trigger of this intestinal Inflammation.

Intestinal inflammation is connected to other extra-intestinal autoimmune inflammations like PSC (as f.ex. the association of PSC with inflammatory bowel disease proves).

Hypothesis: Avoidance of ATIs through a gluten-free diet will reduce intestinal inflammation and thus also the the inflammatory activity in the liver.

Proof of hypothesis:

* Pilot study with n=20 patients with PSC
* Explorative, open-label, mono-centric study
* Inclusion criteria: age 18-65, diagnosed PSC-associated colitis without relevant clinical activity after last coloscopy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed PSC-associated colitis without relevant clinical activity after last coloscopy.

Exclusion Criteria:

* patients with coeliac disease or wheat allergy
* patients with active colitis
* patients already on gluten-free diet
* liver transplanted patients
* patients also diagnosed with autoimmune hepatites (PSC-AIH overlap)
* coloscopy within 2 months before study
* Endoscopic retrograde cholangiopancreatography (ERCP) within 3 months before study
* antibiotics within 3 month before study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Reduction of intestinal inflammatory activity | 2 months
  Expression of pro-inflammatory cytokines in gut mucosa (Sigma)

SECONDARY OUTCOMES:
Inflammatory activity of the liver | 2 months
  alkaline phosphatase (AP)
Reduction of inflammatory cells/markers in the blood | 2 months
  stored blood samples, Pax-Gene
Quality of life | 2 months
  questionnaire
Change of symptoms with change of diet. | 2 months
  questionnaire
Changes in patients microbiota | 2 months (5 months with follow-up)
  stool samples

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liwinski T, Hubener S, Henze L, Hubener P, Heinemann M, Tetzlaff M, Hiller MI, Jagemann B, Surabattula R, Leeming D, Karsdal M, Monguzzi E, Schachschal G, Rosch T, Bang C, Franke A, Lohse AW, Schuppan D, Schramm C. A prospective pilot study of a gluten-free diet for primary sclerosing cholangitis and associated colitis. Aliment Pharmacol Ther. 2023 Jan;57(2):224-236. doi: 10.1111/apt.17256. Epub 2022 Oct 20. PMID 36266939